CLINICAL TRIAL: NCT06973863
Title: A Phase 1a/1b Study Evaluating the Clinical Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-tumor Efficacy of PEP08 as Monotherapy and Combination Therapy in MTAP-Del Advanced or Metastatic Solid Tumors
Brief Title: A Study of PEP08 in Patients With MTAP-Del Advanced or Metastatic Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP08-101
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Solid Tumors; MTAP-deleted Solid Tumors; MTAP Deletion
Keywords: MTAP-del; PRMT5 inhibitor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEP08 monotherapy and expansion in advanced or metastatic solid tumors (Experimental): This arm of the study involves dose escalation to evaluate the tolerability and response of PEP08 monotherapy. Participants in this arm will receive daily dosing and be regularly monitored. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Interventions: Drug: PEP08

INTERVENTIONS:
Drug: PEP08 — PEP08 is an oral, potent, MTA-cooperative PRMT5 inhibitor.

SUMMARY:
This is a first-in-human clinical study of PEP08, a novel cancer therapy being evaluated both as monotherapy and in combination with other treatments in patients with advanced or metastatic solid tumors harboring MTAP deletion.

The study will be conducted in three parts, with Part 1 currently open for enrollment.

The primary objectives of the study are to:

* Evaluate the safety and tolerability of PEP08, PK and PD
* Determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D)
* Assess preliminary signs of anti-tumor activity of PEP08

Key study questions include:

* What is the recommended dose of PEP08 for further development?
* Wht is the tolerable dose of PEP08 when administered alone or in combination?
* Does PEP08 show early evidence of clinical activity in patients with MTAP-deleted tumors?

Participants in the study will:

* Receive PEP08 alone or in combination with another anti-cancer agent, depending on the study part
* Attend regular clinic visits for treatment administration, laboratory assessments, and tumor evaluations
* Be enrolled in one of the following study phases over time:
* - Part 1: Monotherapy dose escalation (currently enrolling).
* - Parts 2 and 3 (monotherapy extension and combination therapy) will be activated in future protocol amendments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults (≥18 years) and sign informed consent before undergoing any study-related procedures.
* Eligible participants must have advanced or metastatic solid tumors that are not treatable with surgery or radiation, and show evidence of MTAP gene homozygous deletion or MTAP protein loss based on tumor tissue analysis.
* Participants must have previously received standard treatment for their cancer type, and either experienced disease progression, be refractory, or be intolerant to such therapies.
* At least one measurable lesion is required, evaluated by standard imaging criteria (RECIST v1.1).
* Good general physical condition (ECOG performance status 0-1 for dose escalation; broader range allowed for other parts).
* Adequate function in key organs.
* Able to swallow oral medication and comply with study requirements.
* Women of childbearing potential and men with reproductive potential must use effective contraception during and after the study.

Exclusion Criteria:

* Recent cancer treatment, immunotherapy, or investigational drugs are not allowed before starting the study.
* Live vaccines received shortly before treatment are not allowed.
* Previous use of drugs with similar mechanisms to the study treatment is not allowed.
* Active or unstable brain or meningeal metastases, unless previously treated and stable without needing local treatment or high-dose steroids.
* History of other cancers within the last 2 years, unless low-risk and treated (e.g., in situ or certain skin cancers).
* Uncontrolled disease-related complications (e.g., abnormal calcium levels, fluid buildup around organs).
* Active HIV, hepatitis B or C infections that are not well-controlled.
* Ongoing serious infections or systemic conditions requiring isolation.
* Significant heart disease, such as recent heart failure, ischemia, or arrhythmias.
* History of severe digestive conditions or surgeries affecting drug absorption.
* Recent major surgery.
* Unresolved serious side effects from prior cancer treatment.
* Currently pregnant or breastfeeding.
* Poorly controlled blood pressure or lung conditions.
* Other serious illnesses (e.g., severe anemia, psychiatric or social issues affecting study compliance).
* Any condition that may pose a safety risk or interfere with the study, as judged by the investigator.
* Known drug or substance abuse that may affect study participation.
* Allergy to the study drug or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AE) | Up to 2 years
Number of Participants Experiencing Serious Adverse Events (SAE) | Up to 2 years
Number of Patients who Experience Dose-Limiting Toxicity | 21 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 6 days
Maximum observed plasma concentration (Cmax) | Up to 6 days
Maximum observed plasma concentration (Cmin) | Up to 6 days
Time to achieve maximal plasma concentration (Tmax) | Up to 6 days
Terminal elimination half-life (t1/2) | Up to 6 days
Objective Response Rate (ORR) per RECIST v1.1 | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Wentworthville, New South Wales, Australia